CLINICAL TRIAL: NCT02305979
Title: Evaluation of Loratadine for Granulocyte-Colony Stimulating Factor Induced Bone Pain in Patients With Hematologic Malignancies
Brief Title: Evaluation of Loratadine for G-CSF Induced Bone Pain in Patients With Hematologic Malignancies
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00030701; CCCWFU 98414 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2014-12-01; First posted 2014-12-03 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma | interventions — Loratadine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment with Loratadine: Treatment with Loratadine
  Interventions: Drug: Loratadine

INTERVENTIONS:
Drug: Loratadine
  Other Names: Claritin

SUMMARY:
The purpose of this project is to assess the efficacy of loratadine in decreasing the incidence and severity of bone pain following G-CSF administration in patients with hematologic malignancies, patients undergoing mobilization of hematopoietic progenitor cells, and patients who have undergone an autologous hematopoietic cell transplant. This is a different patient population than those being assessed in current clinical trials.

DETAILED DESCRIPTION:
Objectives

The primary objective is to determine the incidence of bone pain following G-CSF administration in patients with hematologic malignancies, patients undergoing mobilization of hematopoietic progenitor cells, and patients who have undergone an autologous hematopoietic cell transplant. Incidence will be determined via patient-reported incidence following G-CSF administration.

Secondary objectives include determining the efficacy of loratadine for bone pain prevention as indicated by a decrease in incidence and a decrease in severity (questions 4 and 5 of the survey).

ELIGIBILITY:
Inclusion Criteria:

* Receiving a G-CSF after the institution practice change
* Receiving a G-CSF for one of the following indications:
* Prevention/treatment of neutropenia along with treatment for leukemia or lymphoma
* Mobilization of hematopoietic progenitor cells
* Neutropenia prevention following autologous hematopoietic cell transplant
* Took loratadine per protocol with G-CSF administration
* Completed a survey

Exclusion Criteria:

* Taking daily antihistamines for allergies, asthma, or other indications, not including bone pain
* Taking daily NSAIDs, with the exception of aspirin, for chronic conditions
* Treatment for solid tumor cancers
* Receiving bone modifying agents for bone pain associated with metastatic disease or other chronic conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Wake Forest Baptist Health Hematology and Oncology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Incidence of bone pain following G-CSF administration | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: LeAnne Kennedy, PharmD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States